CLINICAL TRIAL: NCT06019182
Title: Investigations of Individuals With MEHMO Syndrome or eIF2-Pathway Related Conditions
Brief Title: MEHMO Natural History and Biomarkers
Status: Recruiting | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 10001681; 001681-CH
Record Dates: First submitted 2023-08-30; First posted 2023-08-31 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07-24

CONDITIONS: Intellectual Disability; Epilepsy; Hypogonadisms; Microcephaly; Nervous System Malformations; Obesity
Keywords: MEHMO; X-linked MEHMO Syndrome; eIF2-Pathway Related Conditions; EIF2S3
MeSH Terms: conditions — Intellectual Disability; Epilepsy; Microcephaly; Nervous System Malformations; Obesity; MEHMO syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Affected: Individuals who have MEHMO syndrome or eIF2-pathway related conditions 1-week of age or older.
- Carrier: EIF2S3-variant carrier individuals 1-month of age or older.
- Unaffected Non-carrier: Unaffected individuals 1 month of age or older who are 1st degree relative of an affected individual

SUMMARY:
This observational natural history study will follow individuals with MEHMO (Mental disability, Epileptic seizure, Hypopituitarism/Hypogenitalism, Microcephaly, Obesity) syndrome or an eIF2-pathway related disorder, who have symptoms such as intellectual delay, seizures, abnormal hormone and blood sugar levels, and decreased motor skills.

No current treatment for these conditions is available. A major impediment to the testing of potential therapeutic interventions is the lack of well-defined outcome measures. This protocol seeks to identify biochemical and clinical markers to monitor disease progression, and better understand the natural history of these conditions.

Any person diagnosed with MEHMO syndrome or related conditions, who can travel to the NIH Clinical Center can participate in this study.

The study involves:

* General health assessment and evaluation
* Imaging studies
* Laboratory tests
* Collection of blood, urine, spinal fluid, skin biopsy.

DETAILED DESCRIPTION:
Study Description: This is a prospective natural history study of individuals who have MEHMO syndrome or eIF2-pathway related conditions, or who are carriers of EIF2S3-related conditions to generate hypotheses for further understanding of disease pathophysiology, diagnosis, prognosis, management, and treatment. The protocol aims to enroll and follow affected or carrier individuals longitudinally to establish a repository of concurrent evaluations and biomaterials, as well as to enroll unaffected individuals for collection of informative comparable data and samples.

Objectives:

Primary Objective:

Characterize the presentation of MEHMO syndrome and eIF2 pathway related conditions.

Secondary Objectives:

1. Identify disease-reflective fluid biomarkers
2. Develop a disease severity rating scale or classification algorithm
3. Assess tolerability and feasibility of study evaluations
4. Establish a repository of participant data and samples for future research

Endpoints:

Primary Endpoint:

Frequency and time-to-event of signs and symptoms.

Secondary Endpoints:

1. Mean difference of candidate fluid biomarkers level in affected versus carrier versus unaffected individuals
2. Correlation of rating scale or classification algorithm to age, genotype, or other variables
3. Frequency of completed evaluations and reasons for noncompletion

ELIGIBILITY:
* INCLUSION CRITERIA:

To be eligible to participate in this study, an individual must meet the following criteria:

Be >= 1-week of age if affected, or >=1-month of age if unaffected.

For Screening:

1. Have a combination of signs/symptoms suggestive of MEHMO syndrome,

   AND

   no or inconclusive molecular testing.

   OR
2. Be a relative of an individual with MEHMO syndrome/eIF2-related condition and whose genetic may be informative for research.

For Main Study:

1. Have a combination of signs/symptoms suggestive of MEHMO syndrome,

   AND

   disease-associated variant(s) or variant(s) of uncertain significance in one of the eIF2-pathway related genes

   OR
2. Be a relative of an individual with MEHMO syndrome/eIF2-related condition, AND a carrier of the pathogenic or likely pathogenic variant.

   OR
3. Be a non-affected, non-carrier family member of an individual with MEHMO syndrome or an eIF2-pathway related condition.

EXCLUSION CRITERIA:

Any individual who, in the opinion of the Investigators, is unable to comply with the protocol or have medical conditions that would potentially increase the risk of participation will be excluded from participation in this study.

Ages: 1 Week to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Inclusion Criteria: An individual must be > 1-week of age if affected, or > 1-month of age if unaffected. For Screening: Have a combination of signs/symptoms suggestive of MEHMO syndrome, AND no or inconclusive molecular testing. For Main Study: 1. Have a combination of signs/symptoms suggestive of MEHMO syndrome, AND disease-associated variant(s) or variant(s) of uncertain significance in one of the eIF2-pathway related genes OR 2. Be a first-degree relative of an individual with EIF2S3-related MEHMO syndrome, AND a carrier of the pathogenic or likely pathogenic variant. OR 3. Be a non-affected, non-carrier family member of an individual with MEHMO syndrome or an eIF2-pathway related condition. Exclusion Criteria: Any individual who, in the opinion of the Investigators, is unable to comply with the protocol or have medical conditions that would potentially increase the risk of participation.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-10-23 (Actual); Primary Completion 2053-09-01 (Estimated); Study Completion 2053-09-01 (Estimated)

PRIMARY OUTCOMES:
Characterize the presentation of MEHMO syndrome and eIF2-pathway related conditions. | Ongoing
  Frequency and time-to-event of signs and symptoms. These will allow systematic and potentially quantitative measures of disease presentation that can then be operationalized to develop disease rating scale(s) and correlative measures for candidate biomarkers.

SECONDARY OUTCOMES:
Identify disease-reflective fluid biomarkers | Ongoing
  Difference and range of candidate fluid biomarkers level in affected vs. carrier vs. unaffected individuals. Sensitive or specific quantitative markers will allow for improved diagnosis, management, and treatment of MEHMO syndrome or eIF2-pathway related disorders.
Develop a disease severity rating scale or classification algorithm. | Ongoing
  A quantitative rating scale or classification algorithm that reflects other disease aspects will provide a standardized tool for communication amongst all involved in the clinical care and research of MEHMO syndrome or eIF2-pathway related disorders.
Assess tolerability and feasibility of study evaluations. | Ongoing
  Frequency of completed evaluations and reasons for non-completion will inform design of future trials for MEHMO syndrome or eIF2-pathway related disorders.
Characterize EIF2S3-carrier phenotype. | Ongoing
  Frequency and time-to-event of signs and symptoms at disease-relevant intervals will provide a systematic evaluation of EIF2S3- carrier phenotype.
Establish a repository of participant data and samples for future research. | Ongoing
  A repository of concurrently collected participant data and samples for future research will provide resources for future research towards understanding the disease and developing interventions.

CONTACTS AND LOCATIONS:
Overall Officials: An N Dang Do, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
Requests for sharing of relevant IPD for clinical management purpose or directly from the individual participant will be considered on case basis and are not guaranteed to result in sharing of IPD.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_001681-CH.html